CLINICAL TRIAL: NCT02078310
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Oral Dose Escalation for Safety, Tolerability and Pharmacokinetics of ITI-007 in Healthy Geriatric Volunteers and in Geriatric Patients With Dementia.
Brief Title: Study of ITI-007 in Healthy Geriatric Volunteers and in Geriatric Patients With Dementia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: ITI-007-200
Record Dates: First submitted 2014-02-28; First posted 2014-03-05 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2014-11

CONDITIONS: Alzheimer's Disease
Keywords: Dementia,; Healthy; geriatric; volunteers; patients
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — lumateperone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ITI-007 Part 1 (Experimental): Part 1: Healthy geriatric volunteers with multiple oral dose escalation up to and including 20 mg ITI-007
  Interventions: Drug: ITI-007
- Placebo Part 1 (Placebo Comparator): Part 1: Healthy geriatric volunteers with placebo given
  Interventions: Drug: Placebo
- ITI-007 Part 2 (Experimental): Part 2: Geriatric patients with dementia with ITI-007 given
  Interventions: Drug: ITI-007
- Placebo Part 2 (Placebo Comparator): Part 2: Geriatric patients with dementia with placebo given
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ITI-007 — ITI-007 for Part 1
  Arms: ITI-007 Part 1
Drug: Placebo — ITI-007 for Part 1
  Arms: Placebo Part 1
Drug: ITI-007 — ITI-007 for Part 2
  Arms: ITI-007 Part 2
Drug: Placebo — Placebo for Part 2
  Arms: Placebo Part 2

SUMMARY:
A Phase 1b/2, Randomized, Double-blind, Placebo-Controlled, Multiple Oral Dose Escalation Study to Assess Safety, Tolerability and Pharmacokinetics of ITI-007 in Healthy Geriatric Volunteers and in Geriatric Patients with Dementia

ELIGIBILITY:
Inclusion Criteria:

Part 1

* Healthy geriatric volunteers
* MMSE score of >= 26 at screening
* BMI between 19.0 and 40.0 kg/m2 and a minimum body weight of 50 kg at screening

Part 2

* Geriatric patients with a clinical diagnosis of dementia
* MMSE score of < 26 at screening
* BMI between 19.0 and 40.0 kg/m2 and a minimum body weight of 50 kg at screening

Exclusion Criteria:

* Any clinically significant illness within 6 months before screening
* Any history of cancer within last 5 years
* History of Hepatitis B or C infection and elevated ALT, AST or bilirubin above the upper limit of normal level
* Any subject considered to be an imminent danger to themselves or others

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | up to 7 days
  Vital signs, 12-lead ECGs, clinical laboratory testing, and adverse events will be assessed.

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC) | pre-dose and multiple collection points up to 72 h after the last dose

OTHER OUTCOMES:
Exploratory measures of cognitive function | Baseline and up to 7 days
Exploratory measures of agitation | Baseline and up to 7 days
Exploratory measures of subjective sleep | Baseline and up to 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Glendale, California, United States